CLINICAL TRIAL: NCT01292460
Title: A Phase III, Randomized, Double-masked 6-month Trial to Compare the Efficacy and Safety of the Preservative-free Fixed-dose Combination of Tafluprost and Timolol Eye Drops to Those Given Individually in Patients With Open Angle Glaucoma or Ocular Hypertension
Brief Title: Tafluprost-Timolol Preservative-free Fixed Dose Combination (FDC) Superiority Study Against Monotherapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201050
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2011-03

CONDITIONS: Ocular Hypertension; Open-angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — Timolol; tafluprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Preservative-free timolol (Active Comparator)
  Interventions: Drug: Timolol/ FDC/ Placebo/ Tafluprost
- Preservative-free FDC and placebo (Experimental)
  Interventions: Drug: Timolol/ FDC/ Placebo/ Tafluprost
- Preservative-free tafluprost (Active Comparator)
  Interventions: Drug: Timolol/ FDC/ Placebo/ Tafluprost
- Preservative-free FDC (Experimental)
  Interventions: Drug: Timolol/ FDC/ Placebo/ Tafluprost

INTERVENTIONS:
Drug: Timolol/ FDC/ Placebo/ Tafluprost — Prior timolol users: Timolol (administered at 08:00 and 20:00) or FDC of tafluprost and timolol (at 08:00) and Placebo eye drops (at 20:00).
  Prior prostaglandin users: Tafluprost (administered at 08:00) or FDC of tafluprost and timolol (administered at 08:00).

SUMMARY:
The purpose of this study is to compare the efficacy and safety of the preservative-free fixed tafluprost-timolol combination to those of tafluprost and timolol alone. This study will enroll patients who have ocular hypertension or glaucoma and who are using timolol or prostaglandin.

The study medication period is 6 months, but the primary evaluation of efficacy is done at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more
* A diagnosis of ocular hypertension or open-angle glaucoma and prior use of timolol or prostaglandin.
* Meet specific IOP level at visit 1 (screening), visit 2 (run-in) and visit 3 (baseline).
* Meet specific visual acuity score
* Are willing to follow instructions
* Have provided a written informed consent

Exclusion Criteria:

* Females who are pregnant, nursing or planning pregnancy
* IOP of 35 mmHg or greater
* Diagnosis of angle-closure glaucoma or secondary glaucoma other than capsular or pigmentary glaucoma in either eye
* Suspected contraindication or hypersensitivity to study medications tafluprost or timolol (e.g. asthma, low pulse)or to wash-out medication brinzolamide
* Glaucoma filtration surgery or any other ocular surgery (including ocular laser procedures) within 6 months prior to Screening
* Use of contact lenses at Screening or during the study
* Presence of any abnormality or significant illness that could be expected to interfere with the patient safety or study parameters
* Current participation in another clinical trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the average diurnal Intraocular Pressure (IOP) at 3 months | At 3 months

SECONDARY OUTCOMES:
Change from baseline in average diurnal IOP | At 2 and 6 weeks and 6 months
  Change from baseline in the average diurnal IOP at 2 weeks, 6 weeks and 6 months
Change from baseline in timewise IOPs | At 2 weeks, 6 weeks, 3 months and 6 months
  Change from baseline in timewise IOPs (at 8:00, 10:00, 16:00, 20:00)

CONTACTS AND LOCATIONS:
Overall Officials: Auli Ropo, M.D., Study Director — Santen Oy; Hannu Uusitalo, M.D., Prof., Principal Investigator — Tampere University
Locations (2):
- Finland (2):
  - Eye clinic, University Hospital of Kuopio, Kuopio
  - Eye Clinic, University Hospital of Oulu, Oulu

REFERENCES:
- [Derived] Pfeiffer N, Traverso CE, Lorenz K, Saarela V, Liinamaa J, Uusitalo H, Astakhov Y, Boiko E, Ropo A; Preservative-free Tafluprost/Timolol Fixed Combination Study Group. A 6-month study comparing efficacy, safety, and tolerability of the preservative-free fixed combination of tafluprost 0.0015% and timolol 0.5% versus each of its individual preservative-free components. Adv Ther. 2014 Dec;31(12):1228-46. doi: 10.1007/s12325-014-0163-3. Epub 2014 Dec 2. PMID 25447269